CLINICAL TRIAL: NCT05040074
Title: SQ-Kyrin Transcatheter Mitral Valve Repair System Feasibility Study
Brief Title: SQ-Kyrin TMVr FIM Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRP01-001
Record Dates: First submitted 2021-08-12; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Mitral Regurgitation
Keywords: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SQ-Kyrin TMVr Feasibility Study (Experimental): Experimental group is allocated to use the transcatheter edge-to-edge valve repair system of Shanghai Shenqi Medical Technology Co., Ltd.
  Interventions: Device: SQ-Kyrin Transcatheter Edge-to-Edge Valve Repair System

INTERVENTIONS:
Device: SQ-Kyrin Transcatheter Edge-to-Edge Valve Repair System — Transesophageal echocardiography-guided, implantable mitral valve clip repair system

SUMMARY:
A feasibility study to evaluate the effectiveness and safety of the SQ-Kyrin Transcatheter Edge-to-Edge Valve Repair System for the treatment of moderate-to-severe mitral regurgitation in patients with high surgical risk.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm observation, feasibility clinical study that plans to enroll a total of not less than 10 and not more than 30 patients, adopts the post-op immediate technical success rate as the primary endpoint, and uses the all-cause mortality at 30 days post-op, incidence of serious adverse event at 30 days post-op, device success rate at 30 days post-op, and procedural success rate at 30 days post-op as secondary endpoints to evaluate the effectiveness, safety, and feasibility of the Transcatheter Edge-to-Edge Valve Repair System of Shanghai Shenqi Medical Technology Co., Ltd. in clinical use and preliminarily evaluate the product's performance. A phasic study report (for phasic data summary and analysis) will be issued after completion of the 30-day postoperative follow-up to evaluate the effectiveness, safety, and feasibility of the device and apply for clinical studies before official registration and marketing. In the meantime, patients enrolled will continue to be followed up for 6 months and 1-5 years post-op to evaluate the long-term effect of the mitral valve repair system.

ELIGIBILITY:
Inclusion Criteria:

1. Severe mitral valve regurgitation ≥ 3+ (moderate-to-severe mitral regurgitation disease);
2. Patients with high or prohibitive risk for conventional open thoracic surgery as defined by STS risk scoring result; subjects who are judged as not tolerating mitral valve surgery due to STS procedural mortality risk ≥ 8% for mitral valve replacement or presence of any of the following risk factors:

   1. Porcelain aorta or active ascending aortic atheroma
   2. Prior radiation therapy to mediastinum
   3. History of mediastinitis
   4. Left ventricular ejection fraction (LVEF) < 40%
   5. Presence of unobstructed coronary artery bypass graft
   6. History of 2 or more cardiothoracic surgeries
   7. Liver cirrhosis
   8. Other surgical risk factors
3. Degenerated MR patients, or functional MR patients who have received guideline-directed medical therapy (GDMT therapy)
4. Age ≥ 18 years, male or female;
5. Patients who are at extremely high risk or not suitable for conventional mitral valve surgery, as assessed by a multidisciplinary heart team (including at least one cardiac surgeon and one cardiologist);
6. Anatomically suitable for transcatheter mitral valve repair by edge-to-edge technique and can be treated by the SQ-Kyrin device;
7. Patients who can understand the objectives of the trial, volunteer to participate in the study, sign the informed consent form, and are willing to receive related examinations and clinical follow-up.

Exclusion Criteria:

1. History of cardiac and mitral valve surgeries;
2. Infective endocarditis or evidence of active infection;
3. Mitral valve stenosis;
4. Severe uncontrolled coronary artery disease;
5. Pulmonary artery hypertension (systolic pulmonary artery pressure > 70 mmHg);
6. Severe right cardiac insufficiency;
7. LVEF < 30%;
8. Cardiac function of NYHA Class IV;
9. Patient is extremely week to tolerate surgery under general anesthesia, or in a shock state indicating circulatory support;
10. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis;
11. Chronic dialysis;
12. Definite coagulation disorder and severe coagulation system diseases;
13. Clear contraindications for use of anticoagulants;
14. Cerebral stroke or transient ischemic attack in the past 30 days;
15. Any cardiac mass, left ventricular or atrial thrombosis identified by echocardiography;
16. Other valve diseases that requiring surgery or intervention;
17. Severe macrovascular disease requiring surgical treatment;
18. Treatment-naive carotid artery stenosis > 70%;
19. Imaging evidence of inappropriate cardiac and valve anatomy;
20. Known hypersensitivity to contrast media, and nickel-titanium memory alloy products;
21. Severe nervous system disorder compromising the cognitive ability;
22. Life expectancy < 12 months;
23. Severe thorax deformity;
24. Pregnant and lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute procedural success | Immediate postoperative
  Must meet all the four items：1）no procedural mortality; 2）success in delivery and retrieval of the device delivery system; 3）successful deployment and accurate positioning of the device; 4）no emergency surgery or reintervention related to the device or surgical approach

SECONDARY OUTCOMES:
All-cause mortality | 1 month
  Death from any cause
Incidence of serious adverse event(SAE) | 1 month
  If the adverse event meets any of the criteria below, it is regarded as a serious adverse event (SAE): 1) results in death; 2) is life threatening, results in illness or injury; 3) requires inpatient hospitalization or prolongation of existing hospitalization; 4) results in a persistent or significant disability/incapacity; 5) results in a congenital anomaly/birth defect, fetal death, fetal distress; 6) results in medical or surgical intervention to prevent permanent impairment to body structure or a body function; 7) an important medical event that may not result in death, be life-threatening, or require hospitalization but may be considered serious when, based upon appropriate medical judgment, may jeopardize the patient or subject and/or may require intervention to prevent one of the outcomes listed in this definition.
Device success rate | 1 month
  Definition of device success（must meet all the four items） ：1) No procedural mortality or stroke；2) Proper deployment and positioning of the device；3) No emergency surgery or reintervention related to the device or surgical approach；4) The implanted mitral valve repair system achieves the following safety and effectiveness indicators:
  * No evidence of structural or functional abnormality
  * No device-related technical failure or complication
  * Significant functional improvement after valve repair, without significant stenosis (post-op EOA ≥ 1.5 cm2 and transvalvular pressure gradient < 5 mmHg/valve regurgitation ≤ Grade 2+/no device-related hemolysis)
Procedural success rate | 1 month
  Definition of procedural success（must meet the two items）：1) Device success；2) Absence of the following severe complications: death; stroke; life-threatening hemorrhage; severe vascular complications; secondary severe organic heart diseases (e.g.: aortic dissection, left atrium/auricle rupture, left ventricular outflow tract obstruction, etc.); Grade II-III and above renal insufficiency; myocardial infarction or coronary ischemia requiring percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG); severe hypotension, heart failure, respiratory failure requiring use of high-dose vasoactive medications/mechanical acids; any valve-related dysfunctions, including repair device detachment (single or two valve leaflets)/embolism/device-related autologous mitral valve damage/other conditions requiring second intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, PLA, Shenyang, Liaoning, China

DOCUMENTS (1):
  • Study Protocol (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT05040074/Prot_000.pdf